CLINICAL TRIAL: NCT04899752
Title: The Effect of Motivational Interviewing and Clinician Centered Interviewing Based Cardiac Rehabilitation on Core Outcomes
Brief Title: Motivational Interviewing & Clinician Centered Interviewing on Cardiac Rehab
Acronym: MIOPCR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Danielle D Wadsworth, Associate Professor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-512 EP 2011
Record Dates: First submitted 2021-02-08; First posted 2021-05-24 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Cardiac Rehabilitation; Motivational Interviewing
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of three groups.
Who Masked: Participant
Masking Description: Participants will not be award of group assignments as all participants are provided a face-to-face interaction with the provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional OPCR (Experimental): Those who are in the traditional group will discuss topics like medication adherence, physical activity questions, or eating habits without a clear from of autonomy or nonautonomy basis as is currently completed in OPCR. This will occur in a face to face format.
  Interventions: Behavioral: Motivational Interviewing
- OPCR + MI (Experimental): The MI group will be consistent with the spirit of MI and utilize a high autonomy communication style to provide support for behavior change across multiple behaviors. This will occur in a face to face format.
  Interventions: Behavioral: Motivational Interviewing
- OPCR + Clinician centered (Experimental): The OPCR + CC group will participate in low-autonomy face to face interviews. Meaning the communication style will be clinician centered, providing goals to the participants without valuing their input.
  Interventions: Behavioral: Motivational Interviewing

INTERVENTIONS:
Behavioral: Motivational Interviewing — Participants will participate in three different communication styles to determine the effect of MI on cardiac rehab outcome measures.

SUMMARY:
The purpose of this project is to examine the differences in outpatient cardiac rehab (OPCR) core component outcomes on different intervention conditions. Conditions include traditional OPCR (control), OPCR + motivational interviewing (MI) and OPCR + Clinician centered interviews.

DETAILED DESCRIPTION:
Participants who are beginning a OPCR program at a local hospital are eligible for the program. During the standard admission procedures, eligible participants will be provided with a consent from and asked to participate in the study. Participants who provide consent will complete their admission packet. The standard admission packet includes: the Outpatient Fall Assessment Risk, Patient Health Questionnaire (PHQ-9),the Dartmouth Quality of Life, and the Rate Your Plate. In addition participants will complete three additional surveys: the Intrinsic Motivation Inventory (IMI), the FPS, (FACES Pain Scale), and the Brief Resilience Scale (BRS). During their second appointment participants will complete the standard 6 minute walk test which is scheduled at their convenience and the grip strength. Participants will then be randomly assigned to the traditional OPCR, the OPCR + MI, or the OPCR - Clinician centered. Post-testing will include all baseline information as well as information from patients charts (lipid profile, HbA1c, risk factors and family history). Analysis will determine differences in core outcomes between the three groups.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in outpatient cardiac rehab
* Able to complete the paperwork independently

Exclusion Criteria:

* Unable to complete assessments and paperwork independently.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Adherence to CR | 12 weeks
  Differences in the number of sessions attended between groups
6-minute walk | 12 weeks
  Changes in the distance traveled during a 6-minute walk
Rate my plate | 12 weeks
  Changes in heart healthy diet
Dartmouth Quality of Life index | 12 weeks
  Changes in Dartmouth Quality of Life Index. Range is 9-45. Higher score indicates lower quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle D Wadsworth, PhD, Principal Investigator — Auburn University
Locations (1):
- Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
We will not share IPD due to Hippa